CLINICAL TRIAL: NCT05757739
Title: Randomized Controlled Trial (RCT) of Open Debridement Versus Percutaneous Ultrasonic Treatment for Symptomatic Lateral Epicondylitis.
Brief Title: Randomized Controlled Trial (RCT) of Open Debridement Versus Tenex
Acronym: Tenex
Status: Recruiting | Type: Observational
Sponsor: Virtua Health, Inc. (Other)
Collaborators: Dr. Sean Mcmillan (Unknown); Dr. Thomas Plut (Unknown); Dr. Christopher Chung (Unknown); Dr. Raymond Ragland (Unknown); Dr. Nathan Bodin (Unknown)
Responsible Party: Sponsor
Other Study IDs: G23004
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Orthopedic Devices Associated With Misadventures
MeSH Terms: interventions — Guanfacine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tenex — In the Tenex procedure, the surgeon inserts a special needle into the damaged portion of the tendon under ultrasound guidance. Ultrasonic energy vibrates the damaged tissue and it can be suctioned out. This procedure is done with local anesthesia in surgeon's office.

SUMMARY:
Lateral epicondylitis (Tennis Elbow) can cause pain and keep individuals from completing their daily activities and require them to miss work. There are currently different treatment options to address tennis elbow. However surgeons do not know if one is better than the other. This study will compare two treatment options for tennis elbow. Participants will either be treated by Ultrasound-guided Percutaneous Tenotomy Technique or Open Surgical Debridement. Traditional open surgical debridement is a surgical procedure that requires the surgeon to make an incision to remove the damaged tissue. This procedure is done under anesthesia in a surgery center. In the Tenex procedure, the surgeon inserts a special needle into the damaged portion of the tendon under ultrasound guidance. Ultrasonic energy vibrates the damaged tissue and it can be suctioned out. This procedure is done with local anesthesia in surgeon's office.

DETAILED DESCRIPTION:
During the initial screening visit, the physician will obtain your medical history and perform a physical exam. If you pass the screening, you will be randomized into either Ultrasound-guided Percutaneous Tenotomy Technique or Open Surgical Debridement. It will be a 50% chance. It will be compared to flipping a coin.

Once you have been placed in your treatment group, your treatment will be scheduled. You will then undergo your procedure and provided referral for physical therapy. You will also have follow up appointments with your physician to monitor your progress at 3 week(visit 3), 5 weeks (visit 4), 3 months (visit 5) 6 month (visit 6), and 12 month (visit 7) time points. You will also be requested to complete two patient questionnaires about your progress at visits 3-7.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18-70 years of age
* Clinically documented chronic lateral epicondylitis with a minimum of 6 months of persistent elbow pain that impedes daily activities.
* Failed alternative treatment for > 3 months.

Exclusion Criteria:

* Surgical procedure on affected extremity within last six months.
* Dermatological disorder in affected area
* Currently pregnant, confirmed via pregnancy test.
* Blood disorders, autoimmune disorders, disorders requiring immunosuppression, cancer, malignancies, an ongoing infectious disease, or sickle cell or other blood disorders.
* Failed prior surgical procedure on the affected joint.
* No prior effort to treat (stretching, rest, medication) or implementation of external protocol in an effort to improve condition (physical therapy, massage treatment, rehabilitation techniques).

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinically documented chronic lateral epicondylitis with a minimum of 6 months of persistent elbow pain that impedes daily activities.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Background: Ultrasound-guided Percutaneous Tenotomy Technique | 3 months
  Background: Ultrasound-guided Percutaneous Tenotomy Technique

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Virtua Health Inc, Burlington, New Jersey
  - Virtua Health and Wellness, Cherry Hill, New Jersey
  - Virtua Cadiac Testing Center, Moorestown, New Jersey
  - Virtua Hand Surgery, Riverside Park, New Jersey
  - Summit Surgical Center LLC, Voorhees Township, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided